CLINICAL TRIAL: NCT03808454
Title: The Effect of Proprioception of Platelet Rich Plasma for Patients With Ankle Sprain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Shang-Lin Chiang, Director, Department of Rehabilitation, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tri-Service General Hospital
Record Dates: First submitted 2019-01-01; First posted 2019-01-17 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Ankle Sprain 2Nd Degree; Ankle Sprain 3Rd Degree
Keywords: Platelet rich plasma, proprioception, ankle sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelet rich plasma (PRP) (Experimental): PRP injection only
  Interventions: Drug: PRP
- PRP+Rehabilitation (Experimental): PRP injection combined with rehabilitation
  Interventions: Combination Product: PRP+Rehabilitation
- Rehabilitation (Active Comparator): Rehabilitation treatment only
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Drug: PRP — The investigators draw 10cc of blood and concentrate the blood to get the platelet rich plasma
  Arms: Platelet rich plasma (PRP)
Other: Rehabilitation — strengthening ex, posture training,...
  Arms: Rehabilitation
Combination Product: PRP+Rehabilitation — combine PRP and Rehabilitation
  Arms: PRP+Rehabilitation

SUMMARY:
Ankle sprain is a fairly common sports medicine clinic. In Taiwan at least 150,000 to 200,000 people will suffer from ankle sprains every years. Clinicians have been looking for ways to shorten treatment time and reduce discomfort. Platelet Rich Plasma(PRP) is an endogenous therapeutic technology that involved in regenerative medicine due to its potential to stimulate and accelerate tissue healing. PRP can release lots of growth factors like platelet-derived growth factor (PDGF),transforming Growth Factor Beta(TGF-β), vascular endothelial growth factor(VEGF),Epidermal growth factor(EGF) and insulin-like growth factor (IGF). Its use had been based on the theory that increased autologous platelets, that then yield high concentrations of growth factors and other proteins, will lead to increased healing of tendon and soft tissue on a cellular level. In addition, there is no objective evaluation after treatment, so that patients can not provide effective and accurate quantitative feedback. In this study, the investigators divided patients into three groups, respectively, general rehabilitation therapy, autologous PRP injection therapy, autologous PRP injection combined with general rehabilitation therapy.

DETAILED DESCRIPTION:
The investigators divided patients into three groups, respectively, general rehabilitation therapy, autologous PRP injection therapy, autologous PRP injection combined with general rehabilitation therapy randomly. The investigators also use the new ankle proprioception evaluation system and evaluation of clinical function after treatment. It is expected to establish another feasible and rapid treatment method for ankle sprain. Combined with high accuracy ankle body defect evaluation method, it is helpful to design proper treatment and rehabilitation strategy in the future so as to improve the rehabilitation of limbs Coordination and control capabilities.

ELIGIBILITY:
Inclusion Criteria:

* ankle sprain within one months
* Gr II or Gr III ankle sprain (anterior talus fibular ligament)by sonogram proved
* MMSE≥23
* could cooperate the examination of the test

Exclusion Criteria:

* Hemianopsia or hemineglect any brain lesion such as cerebrum of cerebellum involved movement
* cancer victim
* pregnant If needed PRP treatment
* Liver cirrhosis
* Platelet < 150000/UL
* Sepsis, Leukemia
* use anti-coagulation agents
* under hemodialysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
mean of the distance of ankle movement by the force plate system | 10 min
  The proprioception could be evaluated by the parameter of mean of the distance of ankle movement by the force plate system
standard error | 10 min
  evaluated by the parameter of standard error of the distance of ankle movement by the force plate system
coefficient of variance | 10 min
  evaluated by the parameter of coefficient of variance of the distance of ankle movement by the force plate system

SECONDARY OUTCOMES:
Time Up and Go(TUG) | 15 sec
  walking ability
Visual analogues scale (VAS ) | 5 sec
  pain level
AOFAS Ankle-Hindfoot score | 10 min
  function of ankle and foot

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Lin Chiang, PhD, Study Director — Department of rehabiliation,TSGH, Taipei, Taiwan
Locations (1):
- Tri-service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The investigators don't want to share IPD until the investigators publish it.

REFERENCES:
- [Result] L. Laver, M. R. Carmont, M. O. McConkey, E. Palmanovich, E. Yaacobi, G. Mann, et al.,